CLINICAL TRIAL: NCT02071706
Title: Clinical Evaluation of an Integrated PET/MRI System
Acronym: PET/MR_ZURICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114-2013-GES-0010
Record Dates: First submitted 2014-02-23; First posted 2014-02-26 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-01

CONDITIONS: Subjects With Clinical Indication for PET/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm PET/MRI (Other): Single-group evaluation of PET/MRI for diagnostic quality of image
  Interventions: Device: PET/MRI system

INTERVENTIONS:
Device: PET/MRI system — Enrolled subject undergoes PET/MR scan
  Other Names: PET/MRI system inlcudes:; 3T MR750w Magnet; MR750w XRMw Gradient; PET/MRI Body Coil; Photon Detection Ring and PET Detectors; PET/MR Patient Table; PET Electronics (mounted to magnet) and Cables

SUMMARY:
The investigational PET/MRI scanner, including attenuation correction method, is capable of producing diagnostic quality images and appropriate device functionality per user feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a clinical indication for a PET/CT exam
2. Subject must be at least eighteen (18) years of age; and
3. Female subjects that are determined to be non-pregnant by a physician investigator or are demonstrated non-pregnant by negative urine pregnancy test administered within the 24 hour period before PET/CT imaging; and
4. Subject must be able to hear and understand instructions without assistive devices; and
5. Subject must provide written informed consent; and
6. Subject has the necessary mental capacity to understand instructions, and is able to comply with protocol requirements; and
7. Subject is able to remain still for duration of imaging procedure (approximately 60 minutes total for PET/MRI); and
8. Subject must be able to participate in a PET/MR imaging session within 2 hours of concluding their PET/CT exam and within 4 hours of PET radiotracer administration.

Exclusion Criteria:

1. Subjects who have any axial diameter larger than 55 cm; or
2. Subjects with a weight greater than 227 kgs; or
3. Subjects that have metallic/conductive or electrically/magnetically active implants without MR Safe or MR Conditional labeling, with the exception of dental devices/fillings, surgical clips, and surgical staples determined to be safe for MRI scanning by a physician investigator; or
4. Subjects that have implants with MR Unsafe labeling; or
5. Subjects that have implants labeled as MR Conditional by the manufacturer for which the allowable conditions are not expected to be achieved by the MR/PET environment or scan protocol ; or
6. Subjects who have a contraindication to MRI according to the screening policy of the participating site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Duliskovich, Medical Doctor, Study Director — GE Healthcare
Locations (1):
- UniversitätsSpital Zürich, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on January 20, 2014. Last participant enrolled on July 07, 2014 at the Zurich University Hospital site. Subject or participant recruitment was prematurely terminated because the sponsor had determined that sufficient data was collected for regulatory submissions
Pre-assignment Details: Subjects/participants were enrolled in one of three study segments and received a clinically indicated PET/CT exam with radiopharmaceutical injection followed by PET/MRI scanning. Up to two subject datasets (each dataset labelled with unique subject ID) can be collected from one enrolled participant/subject.
Period: Overall Study
Arm/Group | Single-Arm PET/MRI
Started | 62
Completed | 59
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single-Arm PET/MRI
Number analyzed (Participants) | 62
Age, Customized [Count of Participants; unit: Participants] — Patient/participant must be at least 18 years of age. Eligible subjects were allowed to participate up to two times.
  Participants
    Equal to or more than 18 years of age | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Number Usable PET/MRI Image Sets
Description: The number PET/MRI image sets determined usable by a radiologist on a yes/no binary scale
Time Frame: 1 day
Measure: Number; unit: Usable image sets
Arm/Group | Single-Arm PET/MRI
Number analyzed (Participants) | 62
Usable image sets | 70

2. Primary Outcome: Number of Diagnostic Quality Images
Description: Number of images sets deemed diagnostic quality by the investigator
Time Frame: 1 day
Population: PET/MR Scans with qualitative comments
Measure: Number; unit: Image sets
Units Other Than Participants: Number of Image Sets
Arm/Group | Single-Arm PET/MRI
Number analyzed (Participants) | 62
Number analyzed (Number of Image Sets) | 74
Image sets | 67

ADVERSE EVENTS:
Time Frame: approximately 7 months
Description: subject participants were considered to be actively enrolled from the time the subject entered the scan room for their PET/MR procedure to the time the subject left the PET/MR scan room. AE monitoring were conducted starting from the subject participants signing off the informed consent form until the subject participant left the PET/MR scan room
Arm/Group | Single-Arm PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 2/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Arm PET/MRI (N=62)
Warming (Musculoskeletal and connective tissue disorders) | 2 — the two reported AEs (Warming) were considered to be anticipated, mild, and probably device-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less